CLINICAL TRIAL: NCT06975683
Title: Open, Non-comparative, Pilot Study to Evaluate the Safety and Efficacy of Intraovarian Growth Factor-rich Plasma in Patients With Low Ovarian Reserve
Brief Title: Open, Non-comparative Pilot Study to Evaluate the Safety and Efficacy of Intraovarian Plasma Rich in Growth Factors (PRGF) in Patients With Low Ovarian Reserve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: URA-PRGF-01; 2024-514444-87-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-10; First posted 2025-05-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Low Ovarian Reserve
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Intervention Model Description: Quasi-Experimental Study with Pre-Post Comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients starting ovarian stimulation cycle for FIV-ICSI cycle (Experimental)
  Interventions: Biological: Plasma Rich in Growth Factors (PRGF)

INTERVENTIONS:
Biological: Plasma Rich in Growth Factors (PRGF) — On the day of the ovarian puncture of the 1st IVF cycle, intraovarian instillation of plasma rich in growth factors will be performed.

SUMMARY:
The use of plasma rich in growth factors (PRGF) improves ovarian reserve markers and IVF laboratory parameters in women with low ovarian reserve.

Primary objective To compare ovarian reserve markers and IVF-ICSI laboratory results before and after PRGF infusion.

Secondary Objectives

* To compare pre- and post-treatment pregnancy rates.
* To collect complications associated with the application of intraovarian PRGF. General Outline of the Study VISIT 1
* Patient Selection
* Confirm that he/she has all the analyses and variables to be studied.
* Signing of Informed Consent
* Usual IVF protocol (1st IVF cycle) VISIT 2
* Instillation of intraovarian PRGF on the day of the puncture of the 1st IVF cycle in the FJD VISIT 3
* Analytical control at 4 weeks VISIT 4
* Analytical control at 8 weeks VISIT 5
* In case of failure to achieve gestation Start of 2nd cycle of IVF

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing age as defined by the CTFG*.
* Women in group 3 and 4 of the POSEIDON classification for low reserve:
* POSEIDON 3: patients ˂ 35 years of age with decreased ovarian reserve (AMH <1.2 ng/ml, AFC <5).
* POSEIDON 4: patients ≥ 35 years with decreased ovarian reserve (AMH <1.2 ng/ml, AFC <5).
* Patients with at least one ovary.
* Infertility of more than 1 year duration.
* Provision of safe ovarian access on the day of the puncture.
* They agree to participate and to give their written consent.

Exclusion Criteria:

* Have a diagnosis of clinical ovarian insufficiency - Patients with an ongoing pregnancy - Patients with a clinical diagnosis of ovarian failure
* Patients with ongoing pregnancy
* Current or previous IgA deficiency,
* Ovarian failure secondary to identified genetic causes.
* Presence of pelvic adhesions after abdominal surgery.
* Chronic use of aspirin, NSAIDs or anticoagulants.
* Diseases that alter platelet number or function.
* Psychiatric disorder that precludes participation in the study (including active substance abuse or dependence).
* Obesity (BMI ≥ 30).
* Current female smokers (≥ 15 cigarettes per day) - Current smoking (≥ 15 cigarettes per day)
* Patients affected by neoplastic disease
* Severe male factor infertility

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of cycles cancelled pre-puncture | Day 1
Ovarian reserve markers | Day 1 vs visit 4 weeks
Number of cycles cancelled post-puncture | visit 4 weeks and visit 8 weeks
Number of oocytes recovered | visit 4 weeks and visit 8 weeks
Number of MII (metaphase II stage oocyte) on the day of the puncture | visit 2, day of the puncture (from the first day of menstruation, approximately 22 days later)
Number of fertilised oocytes | visit 4 weeks and visit 8 weeks
Number of embryos obtained per EOC (ovarian stimulation) cycle | visit 4 weeks and visit 8 weeks
Number of embryos of good quality (A or B quality according to ASEBIR classification). | visit 4 weeks and visit 8 weeks
Number of frozen embryos | visit 4 weeks and visit 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Jiménez Diaz, Madrid, Spain